CLINICAL TRIAL: NCT02565238
Title: Master Study of the Insertable Cardiac Monitor BioMonitor 2.
Brief Title: BIO.MASTER.BioMonitor 2 Study
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: BA105
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Tachyarrhythmia; Atrial Fibrillation; Syncope
MeSH Terms: conditions — Tachycardia; Atrial Fibrillation; Syncope

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BioMonitor 2 — Implantation of BioMonitor 2

SUMMARY:
The objective of the study is to confirm safety and efficacy of the BioMonitor 2. The data is collected to support the regulatory approval of this product in countries outside the CE region.

ELIGIBILITY:
Inclusion Criteria:

* Patients without history of atrial fibrillation and with an indication for BioMonitor 2 device or paients planned for loop recorded guided AF-therapy management, with either current known and documented paroxysmal atrial fibrillation or with current known and documented persistent atrial fibrillation indicated for an ablation or was ablated within the last four weeks.
* Patient is able to understand the nature of the study and provides written informed consent.
* Patient is able and willing to complete the planned follow-up visits at the investigational site.
* Patient accepts the Home Monitoring® concept.
* Age is ≥ 18 years.

Exclusion Criteria:

* Patients implanted with ICD or pacemaker.
* Patient who is pregnant and/or breast-feeding or who intends to become pregnant during the time of the study will be excluded.
* Life expectancy of less than 6 months.
* Participation in another interventional clinical investigation. Participation in a non-interventional study is permitted.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient collective consists mainly of patients with indications of an insertable cardiac monitor or who are planned for loop recorded guided AF-therapy management. The investigator will select patients who are appropriate for particiation from his general patient population.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Device Effect (SADE)-free rate ≥ 90% related to BioMonitor 2 | 3 month

SECONDARY OUTCOMES:
R-Wave amplitude ≥ 0.3 mV | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Piorkowski, MD, Principal Investigator — Heart Center Dresden, Germany